CLINICAL TRIAL: NCT04767386
Title: Relation Between Near Point of Convergence and Postural Stability in Subjects with Non Specific Cervical Pain
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amina Awad,PhD, Assisted professor, Cairo University
Other Study IDs: P.T. REC/012/001842
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2021-02

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A correlation study was conducted to correlate between the convergence insufficiency and postural stability at three different cervical positions in patients with non-specific cervical pain.

DETAILED DESCRIPTION:
A correlational study was conducted on eighty (male and female) subjects aged between 30-40 years old, presented with chronic NSCP persisted for six months or more, with neck disability index score (NDI) ≥10%, and can possess at least 45° of left and right cervical rotation participated in the study. Convergence insufficiency was evaluated by the near point of conversion (NPOC) rule and postural instability was examined by the Biodex balance system. RESULTS: There was significant positive correlation between (NPOC) and anteroposterior stability index (APSI) at the three cervical positions; neutral, 45° right torsion and 45° left torsion (P>0.05).

ELIGIBILITY:
Inclusion Criteria:

* Age from 30 to 40 years.
* Chronic cervical pain ( 6 to18 months ago).
* Neck Disability Index (NDI) score ≥10%),
* Move 45° of cervical rotation to both the left and right.

Exclusion Criteria:

-Neuromuscular or musculoskeletal disorders.

Ages: 30 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Egyptian subjects
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Stability index | during the procedure
  Antero-posterior and mediolateral stability index
The near point of convergence (NPOC) | during the procedure
  The near point of convergence (NPOC) measured by NPOC rule
The CROM | during the procedure
  cervical flexion, extension, rotation and lateral flexion

CONTACTS AND LOCATIONS:
Overall Officials: Wael Shendy, PhD, Study Director — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Cairo Governorate, Egypt